CLINICAL TRIAL: NCT01969240
Title: Shared Decision Making in the Emergency Department: The Chest Pain Choice Trial
Brief Title: Shared Decision Making in the Emergency Department: Chest Pain Choice Trial
Acronym: CPC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Indiana University (Other); University of California, Davis (Other); Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Erik P. Hess, MD, MSc, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 13-001359
Record Dates: First submitted 2013-10-17; First posted 2013-10-25 (Estimated); Results first posted 2018-08-06 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2017-11

CONDITIONS: Chest Pain; Acute Coronary Syndrome
Keywords: Chest Pain; Decision Aid; Acute Coronary Syndrome; Cardiac; Emergency Department; Cardiac Testing; Healthcare Utilization; Patient Centered Outcomes; Shared Decision Making; Unnecessary hospital admissions
MeSH Terms: conditions — Chest Pain; Acute Coronary Syndrome; Emergencies

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chest Pain Choice Decision Aid (Active Comparator): Patients randomized to the decision aid arm.
  Interventions: Other: Chest Pain Choice Decision Aid
- Usual Care (No Intervention): Patients randomized to the usual care arm (no decision aid used)

INTERVENTIONS:
Other: Chest Pain Choice Decision Aid — The clinician will review the decision aid with the patient. The decision aid will be used as a tool to facilitate discussion and educate the patient regarding the rationale for their evaluation up to that point in the emergency department visit and their individual risk for a heart attack or pre-heart attack. The clinician will provide the patient with management options consistent with both the patient's values and preferences and the clinician's level of comfort.
  Other Names: CPC DA
  Arms: Chest Pain Choice Decision Aid

SUMMARY:
Our long-term goal is to promote evidence-based patient-centered evaluation in the acute setting to more closely tailor testing to disease risk. To compare the use of risk stratification tools with usual clinical approaches to treatment selection or administration, we propose the following:

1. Test if Chest Pain Choice safely improves validated patient-centered outcome measures in a pragmatic parallel patient randomized trial.

   Hypothesis: The intervention will significantly increase patient knowledge, engagement, and satisfaction with no increase in adverse events.
2. Test if the decision aid has an effect on healthcare utilization within 30 days after enrollment.

Hypothesis: The intervention will significantly reduce the rate of hospital admission, rate of cardiac testing, and total healthcare utilization.

ELIGIBILITY:
Inclusion Criteria:

1. 18+ years of age (at least 18).
2. Admitted to emergency department for chest pain.
3. Being considered by the treating clinician for admission for cardiac testing.

Exclusion Criteria:

1. Ischemic changes on the electrocardiogram not known to be old as determined by the treating clinician in real time.
2. Elevated cardiac troponin (cTn) above the 99th percentile reference limit.
3. Known coronary artery disease as defined by consensus guidelines on risk stratification studies for emergency department patients with potential acute coronary syndrome (≥ 50% stenosis on cardiac catheterization; prior electrocardiographic changes indicative of ischemia, e.g., ST-segment depression, T-wave inversion, or left bundle branch block; perfusion defects or wall motion abnormalities on previous exercise, pharmacological, or rest imaging studies; previous documentation of acute myocardial infarction; or, if no records are available, patient self-report of coronary artery disease).
4. Cocaine use within the previous 72 hours by clinician history.
5. Pregnancy.
6. Referral to the emergency department by a personal physician for admission.
7. Patients who indicate that a hospital different than the site hospital is his or her "hospital of choice" in the event of a return emergency department visit.
8. Patients undergoing medical clearance for a detox center or any involuntary court or magistrate order.
9. Homelessness, out-of-town residence or other condition known to preclude follow-up.
10. Patients in police custody or currently incarcerated individuals.
11. Patients who have, in their clinician's best judgment, major communication barriers such as visual or hearing impairment or dementia that would compromise their ability to give written informed consent (or use the decision aid).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 898 (Actual)
Dates: Start 2013-10; Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erik Hess, MD, MSc, Principal Investigator — Mayo Clinic, Rochester, MN
Locations (5):
- United States (5):
  - University of California, Davis, Sacramento, California
  - Mayo Clinic, Jacksonville, Florida
  - Indiana University Hospital: IU, Indianapolis, Indiana
  - Mayo Clinic, Rochester, Minnesota
  - Thomas Jefferson University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
A link to the pre-test probability web tool and the Chest Pain Choice decision aid (DA) can be accessed at the Mayo Clinic Shared Decision Making National Resource Center at http://shareddecisions.mayoclinic.org/decision-aid-information/chest-pain-choice-decision-aid/. De-identified patient level data and statistical code can be requested from the corresponding author at hess.erik@mayo.edu and provided to investigators who agree to adhere to a signed research data use agreement with the Mayo Clinic after 12/31/2017.

REFERENCES:
- [Derived] Hess EP, Hollander JE, Schaffer JT, Kline JA, Torres CA, Diercks DB, Jones R, Owen KP, Meisel ZF, Demers M, Leblanc A, Shah ND, Inselman J, Herrin J, Castaneda-Guarderas A, Montori VM. Shared decision making in patients with low risk chest pain: prospective randomized pragmatic trial. BMJ. 2016 Dec 5;355:i6165. doi: 10.1136/bmj.i6165. PMID 27919865
- [Derived] Anderson RT, Montori VM, Shah ND, Ting HH, Pencille LJ, Demers M, Kline JA, Diercks DB, Hollander JE, Torres CA, Schaffer JT, Herrin J, Branda M, Leblanc A, Hess EP. Effectiveness of the Chest Pain Choice decision aid in emergency department patients with low-risk chest pain: study protocol for a multicenter randomized trial. Trials. 2014 May 10;15:166. doi: 10.1186/1745-6215-15-166. PMID 24884807

RESULTS

PARTICIPANT FLOW:
Groups:
- Chest Pain Choice Decision Aid: Patients randomized to the decision aid arm
  Chest Pain Choice Decision Aid: The clinician will review the decision aid with the patient. The decision aid will be used as a tool to facilitate discussion and educate the patient regarding the rationale for their evaluation up to that point in the ED visit and their individual risk for a heart attack or pre-heart attack. The clinician will provide the patient with management options consistent with both the patient's values and preferences and the clinician's level of comfort.
Period: Overall Study
Arm/Group | Chest Pain Choice Decision Aid | Usual Care
Started | 451 | 447
Completed | 451 | 447
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients presenting to a participating emergency department for evaluation of chest pain.
Groups:
- Chest Pain Choice Decision Aid: Patients randomized to the decision aid arm.
  Chest Pain Choice Decision Aid: The clinician will review the decision aid with the patient. The decision aid will be used as a tool to facilitate discussion and educate the patient regarding the rationale for their evaluation up to that point in the ED visit and their individual risk for a heart attack or pre-heart attack. The clinician will provide the patient with management options consistent with both the patient's values and preferences and the clinician's level of comfort.
- Total: Total of all reporting groups
Arm/Group | Chest Pain Choice Decision Aid | Usual Care | Total
Number analyzed (Participants) | 451 | 447 | 898
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.0 (15.0) | 50.6 (14.1) | 50.3 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 274 | 260 | 534
  Male | 177 | 187 | 364
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 4 | 8
  Asian | 6 | 9 | 15
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 155 | 154 | 309
  White | 262 | 269 | 531
  More than one race | 22 | 11 | 33
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 451 | 447 | 898

OUTCOME MEASURES:

1. Primary Outcome: Test if Chest Pain Choice Safely Improves Patient Knowledge.
Description: Patient knowledge was measured by immediate post-visit survey that included 8 questions about the patient's risk for acute coronary syndrome and the available management options.
Time Frame: Directly following intervention (on day 1)
Measure: Mean (Standard Deviation); unit: number of questions correct
Arm/Group | Chest Pain Choice Decision Aid | Usual Care
Number analyzed (Participants) | 451 | 447
number of questions correct | 4.2 (1.5) | 3.6 (1.5)
Statistical Analysis 1: Comparison: Chest Pain Choice Decision Aid vs Usual Care; Test type: Superiority; Mean Difference (Final Values) = 0.66, 95% CI 2-sided [0.46 to 0.86]

2. Secondary Outcome: Test if the Decision Aid Has an Effect on Healthcare Utilization Within 30 Days After Enrollment.
Description: We will measure the effect of the decision aid on the frequency of hospital admission and cardiac testing within 30 days of enrollment.
Time Frame: Within 30 days of study enrollment
Measure: Number; unit: participants
Arm/Group | Chest Pain Choice Decision Aid | Usual Care
Number analyzed (Participants) | 451 | 447
participants
  Admitted to the hospital | 22 | 22
  Cardiac stress testing | 172 | 204
Statistical Analysis 1: Comparison: Chest Pain Choice Decision Aid vs Usual Care; Test type: Superiority; p < 0.013, t-test, 2 sided; The a-priori significance level was 0.05

3. Secondary Outcome: Test if the Decision Aid Safely Improves Patient Engagement.
Description: 1) Patient engagement in the decision-making process as measured by the OPTION scale. The OPTION scale is composed of 12 items with a value of 0-4; they are summed, divided by 48, and then multiplied by 100. Scores range from 0-100, where higher scores are reflective of higher levels of patient engagement.
Time Frame: Immediately after the intervention (on day 1)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Chest Pain Choice Decision Aid | Usual Care
Number analyzed (Participants) | 451 | 447
units on a scale | 18.3 (9.4) | 7.9 (5.4)
Statistical Analysis 1: Comparison: Chest Pain Choice Decision Aid vs Usual Care; Test type: Superiority; Mean Difference (Final Values) = 10.3, 95% CI 2-sided [9.1 to 11.5]

4. Secondary Outcome: Major Adverse Cardiac Event (MACE)
Description: A MACE was defined as acute myocardial infarction, death due to a cardiac or unknown cause, emergency revascularization, ventricular arrhythmia, or cardiogenic shock.
Time Frame: within 30 days of enrollment
Measure: Number; unit: participants
Arm/Group | Chest Pain Choice Decision Aid | Usual Care
Number analyzed (Participants) | 451 | 447
participants | 1 | 0
Statistical Analysis 1: Comparison: Chest Pain Choice Decision Aid vs Usual Care; Test type: Superiority; p = 0.998, Regression, Logistic

5. Secondary Outcome: Total Testing Within 45 Days (a Component of Healthcare Utilization)
Description: In addition to measuring the effect of the decision aid on the frequency of hospital admission and cardiac testing within 30 days, we measured the total number of tests of any type within 45 days. Although we pre-specified 30-day healthcare utilization, on further discussion among the investigative team the consensus was that we collected utilization data out to 45 days and reporting testing utilization at 45 days will provide more robust results.
Time Frame: 45 days
Measure: Mean (Standard Deviation); unit: number of tests obtained
Arm/Group | Chest Pain Choice Decision Aid | Usual Care
Number analyzed (Participants) | 451 | 447
number of tests obtained | 13.3 (6.9) | 14.7 (7.7)
Statistical Analysis 1: Comparison: Chest Pain Choice Decision Aid vs Usual Care; Test type: Superiority; p < 0.001, negative binomial model

6. Secondary Outcome: Decisional Conflict
Description: Decisional conflict, which represents the degree of uncertainty patients experience related to feeling uninformed about the management options, is measured by the decisional conflict scale. The decisional conflict scale includes 16 items that are scored from 0-4; the items are summed, divided by 16, and then multiplied by 25. The scale is from 0-100, where higher scores are reflective of increased patient uncertainty about the choice.
Time Frame: Immediately after the visit (day 1)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Chest Pain Choice Decision Aid | Usual Care
Number analyzed (Participants) | 451 | 447
units on a scale | 43.5 (15.3) | 46.4 (14.8)
Statistical Analysis 1: Comparison: Chest Pain Choice Decision Aid vs Usual Care; Test type: Superiority; Mean Difference (Final Values) = -2.9, 95% CI 2-sided [-4.8 to -0.90]

7. Secondary Outcome: Physician Trust
Description: The trust in physician scale consists of 9 items scored from 1-5; the items are subtracted by 1, summed, divided by 9, and then multiplied by 25. The scale ranges from 0-100, where higher values are reflective of higher levels of patient trust in their physician.
Time Frame: Immediately after the visit (day 1)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Chest Pain Choice Decision Aid | Usual Care
Number analyzed (Participants) | 451 | 447
units on a scale | 89.5 (13.4) | 87.7 (16.0)
Statistical Analysis 1: Comparison: Chest Pain Choice Decision Aid vs Usual Care; Test type: Superiority; Median Difference (Final Values) = 1.7, 95% CI 2-sided [-0.2 to 3.6]

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Chest Pain Choice Decision Aid | Usual Care
Serious Adverse Events (participants affected / at risk) | 1/451 | 0/447
Other Adverse Events (participants affected / at risk) | 4/451 | 1/447
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chest Pain Choice Decision Aid (N=451) | Usual Care (N=447)
Major adverse cardiac event (Cardiac disorders) | 1 (1) | 0 (0) — This intervention patient was admitted to the hospital, had a negative nuclear perfusion stress test, was discharged, and returned to the ED within 30 days with a NSTEMI. The DSMB classified this event as not related to the intervention.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chest Pain Choice Decision Aid (N=451) | Usual Care (N=447)
Acute myocardial infarction (Cardiac disorders) | 4 (4) | 1 (1) — These patients were appropriately diagnosed with an acute myocardial infarction during their index visit to the emergency department.

LIMITATIONS AND CAVEATS:
The study had 78% power to detect a 5% difference in major adverse cardiac event (MACE) rate between study arms, using a 1-sided non-inferiority test with an alpha of 0.05.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No